CLINICAL TRIAL: NCT06587178
Title: Semi-elemental Versus Polymeric Exclusive Enteral Nutrition in the Preoperative Optimization for Patients with Crohn's Disease: a Randomized Controlled Trial
Brief Title: Semi-elemental Versus Polymeric EEN in the Preoperative Optimization for Patients with CD
Acronym: SEPEN-CD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Zhou (Other)
Responsible Party: Sponsor-Investigator, Wei Zhou, Clinical Professor, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210323-11
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease; Nutrition Disorders; Surgery
Keywords: Crohn's disease; Exclusive enteral nutrition; surgery
MeSH Terms: conditions — Crohn Disease; Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SED patient (Experimental): SED patients who received semi-elemental exclusive enteral nutrition.
  Interventions: Dietary Supplement: peptison liquid
- PD patient (Placebo Comparator): PD patients who received polymeric exclusive enteral nutrition.
  Interventions: Dietary Supplement: Enteral nutritional suspension

INTERVENTIONS:
Dietary Supplement: peptison liquid — CD patients requiring bowel resection and preoperative EEN were randomized to receive peptison liquid for 6 weeks.
  Other Names: Nutricia, Amsterdam, Netherlands
  Arms: SED patient
Dietary Supplement: Enteral nutritional suspension — CD patients requiring bowel resection and preoperative EEN were randomized to receive enteral nutritional suspension for 6 weeks.
  Other Names: Nutricia, Amsterdam, Netherlands
  Arms: PD patient

SUMMARY:
Growing evidence has shown that exclusive enteral nutrition (EEN) plays an important role in the preoperative optimization for patients with Crohn's disease (CD). However, the efficacy and safety of different types of enteral feeds including semi-elemental and polymeric enteral nutrition on CD have not been investigated. The aim of this study was to compare the role of semi-elemental and polymeric enteral nutrition on CD.

DETAILED DESCRIPTION:
Growing evidence has shown that exclusive enteral nutrition (EEN) plays an important role in the preoperative optimization for patients with Crohn's disease (CD). However, the efficacy and safety of different types of enteral feeds including semi-elemental and polymeric enteral nutrition on CD have not been investigated. The aim of this study was to compare the role of semi-elemental and polymeric enteral nutrition on CD. The primary outcome: the reduction rate of CRP/ALB after exclusive enteral nutrition in Crohn's disease. The other outcomes: (1) the changes in Crohn's disease activity index; (2) the tolerance of enteral nutrition; (3) the changes in body mass index; (4) postoperative complications and the incidence of stoma; (5) the rate of surgery; (6) other adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. elective bowel resection for Crohn's disease;
2. preoperative diagnosis of Crohn's disease;
3. age between 18 to 65 years old;
4. malnutrition;
5. the Crohn's disease activity index over 150;
6. nasal feeding.

Exclusion Criteria:

1. emergency surgery;
2. preoperative exclusive enteral nutrition before three months;
3. can not tolerate enteral nutrition;
4. less than 6 weeks of exclusive enteral nutrition;
5. preoperative corticosteroids within 3 months;
6. history of gastrointestinal surgery;
7. isolated colon disease;
8. metabolic disease (diabetes, hyperthyroidism).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The change of CRP/ALB level | 6 weeks
  The ratio of C-reactive protein to albumin level changed after exclusive enteral nutrition.

SECONDARY OUTCOMES:
BMI | 6 weeks
  The BMI level changed after exclusive enteral nutrition.
CDAI | 6 weeks
  Crohn's disease activity index, from 0 to 600, the higher index shows more serious of CD.
postoperative complications | 6 weeks
  The incidence of postoperative complications in two groups.
adverse reaction | 6 weeks
  The incidence of adverse reaction during exclusive enteral nutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Xiujun Cai, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Wei Zhou, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data can be available from the email (gxlmed@zju.edu.cn)